CLINICAL TRIAL: NCT03411993
Title: Prevalence of Rheumatic Heart Disease in Pregnancy Among a Population of Antenatal Patients at a Tertiary Care Institution in Western Kenya
Brief Title: Prevalence of Rheumatic Heart Disease Among Pregnant Women in Kenya
Status: Completed | Type: Observational
Sponsor: Moi University (Other)
Collaborators: Moi Teaching and Referral Hospital (Other); Mount Sinai Hospital, Canada (Other); Duke University (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Principal Investigator, Astrid Christoffersen-Deb, Visiting Lecturer, Moi University
Other Study IDs: UMoi4
Record Dates: First submitted 2018-01-17; First posted 2018-01-26 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Cardiac Disease; Pregnancy Related
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Focused cardiac echography — All pregnant women attending antenatal care will be eligible to undergo focused cardiac echo to identify underlying cardiac disease

SUMMARY:
There is currently no routine screening for cardiac disease for pregnant women in areas of high prevalence. This study will aim to determine the point prevalence of cardiac disease in women presenting for antenatal care at Moi Teaching and Referral Hospital. More specifically, it will aim to use focused echocardiography as a screening tool to determine the prevalence of cardiac disease among pregnant women attending MTRH antenatal clinic.

DETAILED DESCRIPTION:
Rheumatic heart disease (RHD) in pregnancy can be associated with severe maternal and neonatal morbidity and mortality. Early identification of these women and referral to specialized, multi-disciplinary care is essential. Overall, studies on RHD prevalence are lacking in sub-Saharan countries and a significant gap in the literature exists for the prospective assessment of disease in the context of pregnancy. At Moi Teaching and Referral Hospital, there are an estimated 3-4 cases per month of women presenting with acute exacerbations of either known or newly diagnosed cardiac disease. These women are often the most challenging clinically and emotionally for the reproductive health team to manage, and contribute to a significant number of the 2-3 maternal deaths per month at MTRH. There is currently no routine screening for cardiac disease in the MTRH antenatal clinics. This study will aim to determine the point prevalence of cardiac disease in women presenting for antenatal care at Moi Teaching and Referral Hospital. More specifically, it will aim to: 1. Use focused echocardiography as a screening tool to evaluate cardiac structure and function; 2. Use focused echocardiography as a screening tool to determine the prevalence of cardiac disease among pregnant women attending MTRH antenatal clinic.; 3. Determine the proportion of pregnant women with cardiac disease who endorse clinical symptoms as a potential means to develop a screening tool; 4. Promote a case-finding culture for cardiac disease in pregnancy

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at any gestational age
* capable to give informed consent

Exclusion Criteria:

* medically unstable: any condition or complication resulting from or independent of pregnancy that necessitates urgent care or that precludes full and informed consent process

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All pregnant women attending the antenatal clinic at Moi Teaching and Referral Hospital. This clinic serves approximately 750 women per month. These women draw from urban, peri-urban and rural areas. As this is a public hospital, income and education levels are low.
Sampling Method: Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Cardiac disease | through study completion, an average of 3 months
  Point prevalence of cardiac lesions identifiable by cardiac echo

CONTACTS AND LOCATIONS:
Overall Officials: John Snelgrove, MD, Principal Investigator — University of Toronto
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No